CLINICAL TRIAL: NCT02078427
Title: ADVATE/ ADYNOVI Hemophilia A Outcome Database
Brief Title: ADVATE/ ADYNOVI Hemophilia A Outcome Database (AHEAD)
Acronym: AHEAD
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 061001
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAX 855

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- rAHF-PFM: Participants treated with rAHF-PFM alone
  Interventions: Biological: ADVATE
- rAHF-PEG: Participants treated with rAHF-PEG alone
  Interventions: Biological: ADYNOVI
- rAHF-PFM then rAHF-PEG: Participants treated with rAHF-PFM and subsequently switched to rAHF-PEG
  Interventions: Biological: ADVATE; Biological: ADYNOVI

INTERVENTIONS:
Biological: ADVATE — Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method
  Other Names: octocog alfa; rAHF-PFM
  Groups: rAHF-PFM; rAHF-PFM then rAHF-PEG
Biological: ADYNOVI — Antihemophilic Factor (Recombinant) Pegylated
  Other Names: rurioctocog alfa pegol; rAHF-PEG
  Groups: rAHF-PEG; rAHF-PFM then rAHF-PEG

SUMMARY:
The purpose of the study is to document the natural history of hemophilia A disease and long-term outcomes in terms of effectiveness, safety and quality of life in participants receiving Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM) or Antihemophilic Factor (Recombinant) - Pegylated (rAHF-PEG) in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Participant has hemophilia A {FVIII lesser than or equal to (<=)5%}
* Participant is prescribed Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM) or Antihemophilic Factor (Recombinant) - Pegylated (rAHF-PEG) by the treating physician
* Participant or participant's legally authorized representative provides informed consent

Exclusion Criteria:

* Participant has known hypersensitivity to the active substance or any of the excipients
* Participant has known allergic reaction to mouse or hamster proteins
* Participant has participated in another clinical study involving an investigational product (IP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving another FVIII concentrate or device during the course of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include male and female participants of any race and age who have a diagnosis of hemophilia A (Factor VIII (FVIII) =5%). Participants must have been prescribed rAHF-PFM or rAHF-PEG for the management of hemophilia A by the treating physician prior to the decision to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Joint Health Outcomes - Assessed by Physical Exam Using Only the Pain, Bleeding, and Physical Exam Parameters of the Gilbert Scale | Up to approximately 12 years
  The World Federation of Hemophilia developed a musculoskeletal evaluation system, commonly referred to as the Gilbert test, to measure hemophilia joint health status.The Gilbert test needs to be performed in the absence of acute bleed, acute pain, and acute inflammation into the evaluated joint. Four parameters are used in each Gilbert test: pain (score: 0-3), bleeding (score: 0-3), physical exam (score: 0-12), and X-ray evaluation (score: 0-13) Scores of 0, represent no pain, no bleeding, no physical exam issues, and/or no x-ray issues. Higher scores for each of these categories represents worsening conditions.

SECONDARY OUTCOMES:
Annualized Bleed Rate, All Joints | Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  The annualized bleed rate for all joints will be calculated per participant and summarized over the set of available participants with a minimum observation period of 90 days per treatment regimen.
Annualized Bleed Rate, All Bleeds | Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  The annualized bleed rate for all bleeds will be calculated per participant and summarized over the set of available participants.with a minimum observation period of 90 days per treatment regimen.
Annualized bleed rate, pre-existing target joints at baseline | Screening visit; Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  The annualized bleed rate for pre-existing target joints at baseline will be calculated per participant and summarized over the set of available participants with a minimum observation period of 90 days per treatment regimen.
Incidence of New Target Joints | Screening visit; Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  The incidence of new target joints will be calculated as the total number of new target joints in all participants divided by the total number of observation days.
Status of joint health by X-ray by Pettersson scale | Screening visit; Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit.
  The status of joint health by X-ray by Pettersson score will be summarized for each observational year.
Status of Joint Health by Magnetic Resonance Imaging (MRI) Scoring System- Using The Lund Scoring System (LSS) | Screening visit; Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  LSS score format= A(e:s:h). Sum of values for Subchondral Cyst (score: 1-6), irregularity/erosion of Subchondral Cortex (score: 1-4), and Chondral Destruction (score: 1-6) gives value for the A component of score. e, s, h components represent effusion/hemarthrosis, hypertrophic synovial, & hemosiderin deposition (score: 0-4 for each). Max. score is 16(4:4:4).
  Subchondral Cyst:
  * ≥1 bone
  * ≥2 bones
  * >3 cysts in ≥1 bone
  * >3 cysts ≥2 bones
  * Largest size >4 mm: ≥1 bone
  * Largest size >4 mm: ≥2 bones
  Subchondral Cortex
  * ≥1 bone
  * ≥2 bones
  * Involve > half joint surface: ≥1 bone
  * Involve > half of joint surface: ≥2 bones
  Chondral Destruction
  * ≥1 bone
  * ≥2 bones
  * Full thickness defect (FTD): ≥1 bone
  * FTD: ≥2 bones
  * FTD involves >1/3 of joint surface: ≥1 bone
  * FTD involves >1/3 of joint surface: ≥2 bones
  Effusion/hemarthrosis (e): Hypertrophic synovial (s): Hemosiderin (h): (0-4 for each):
  * 0 absent
  * 1 equivocal
  * 2 small
  * 3 moderate
  * 4 large
Status of joint health using the Hemophilia Joint Health Score (HJHS) | Screening visit; Annual/Interval visits:- Up to 8 years if rAHF-PFM alone- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  The International Prophylaxis Study Group (IPSG) developed a scoring system for musculoskeletal evaluation, the HJHS, optimized for use in children with no or minimal joint disease.
  The HJHS includes the following parameters: swelling, duration of swelling, muscle atrophy, joint pain, crepitus on motion, flexion loss, extension loss, strength and global gait.
Overall effectiveness assessment for prophylaxis therapy | Annual/Interval visits:- Up to 8 years if rAHF-PFM alone;- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years;- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  * Excellent: Same or lower breakthrough bleed rate (BBR) within last 12 months (M) compared with prior prophylaxis; if participant did not receive prior prophylaxis with rAHF-PFM, rAHF-PEG or other Factor VIII (FVIII), same or better than expected outcome according to investigator's expectation
  * Good: Minor increase in BBR within last 12M compared with prior prophylaxis; if participant did not receive prophylaxis with rAHF-PFM, rAHF-PEG or other FVIII, slightly less than expected outcome according to investigator's expectation
  * Fair: Moderate increase in BBR in last 12M compared with prior prophylaxis; if participant did not receive prophylaxis with rAHF-PFM, rAHF-PEG or other FVIII, somewhat less than expected outcome according to investigator's expectation
  * Poor: Significant increase in BBR in the 12M compared with prior prophylaxis; if participant did not receive prophylaxis with rAHF-PFM, rAHF-PEG or other FVIII, little to no benefit according to investigator's expectation
Compliance with the dosing prescribed and its relationship with effectiveness | Annual/Interval visits:- Up to 8 years if rAHF-PFM alone;- Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years;- Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  Evaluation of patients´ compliance to prescribed prophylactic treatment will be performed by the treating physician. Compliance will be categorized according to a 4-point table (Highly compliant, Fairly compliant, Moderately compliant, Poorly compliant)
Overall effectiveness assessment for on-demand treatment | Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  * Excellent: Bleed episodes typically respond to same or fewer number of infusion and same or lower dose as compared with previous on-demand treatment or investigator's expectation
  * Good: Most bleed episodes typically respond to same number of infusion and dose but some require more infusions or higher dose as compared with previous on-demand treatment or investigator's expectation
  * Fair: Bleed episodes typically require more infusions and/or higher dose than expected as compared with previous on-demand treatment or investigator's expectation
  * Poor: Bleed episodes routinely fail to respond to same number of infusion and dose and require additional or different factor concentrate for hemostatic control as compared with previous on-demand treatment or investigator's expectation
Global effectiveness assessment for on-demand treatment | Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  * Excellent: Full relief of pain and cessation of bleeding as evidenced by objective signs (e.g., swelling, tenderness, irritability, inconsolability, and decreased range of motion in the case of musculoskeletal hemorrhage) within approximately 8 hours of a single infusion. No additional infusion is required for the control of bleeding. Administration of further infusions to maintain hemostasis would not affect this scoring.
  * Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after the infusion. Possibly requires more than 1 infusion for complete resolution.
  * Fair: Probable or slight relief of pain and slight improvement in signs of bleeding within approximately 8 hours after the infusion. Requires more than 1 infusion for complete resolution.
  * Poor: No improvement or condition worsens.
Number of rAHF-PFM or rAHF-PEG units required for bleed cessation | Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM) Antihemophilic Factor (Recombinant) - Pegylated (rAHF-PEG)
Number of rAHF-PFM or rAHF-PEG infusions required for bleed cessation | Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
  Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method (rAHF-PFM) Antihemophilic Factor (Recombinant) - Pegylated (rAHF-PEG)
Incidence of target joint intervention, including surgery, radiosynovectomy, and chemosynovectomy | Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; and Termination visit
Incidence of pseudo tumor development | Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
Quality of Life: HAL questionnaire - for adult patients | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The the lHAL measures activities involving the upper extremities, basic activities involving ower extremities and complex activities involving the lower extremities as well as an overall physical activity score for adults.
Quality of Life: SF-12v2 questionnaire - for adult patients | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The SF-12v2 measures generic health-related quality of life for adults.
Quality of Life: EQ-5D questionnaire - for adult patients | Enrollment visit;Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The EQ-5D measures health utility in adult participants.
Quality of Life: PedHAL questionnaire - for pediatric patients | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The PedHAL measures activities involving the upper extremities, basic activities involving the lower extremities and complex activities involving the lower extremities as well as an overall physical activity score for children.
  For participants 4-13 years of age:
  - PedHAL (parent version)
  For participants 14-17 years of age:
  - PedHAL (child version)
Quality of Life: SF-10 questionnaire - for pediatric patients | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The SF-10 measures generic health-related quality of life for children and is parent-completed.
Quality of Life: EQ-5D (14 and up) questionnaire - for pediatric patients | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The EQ-5D measures health utility in subjects aged 14 and up.
Chronic pain associated with hemophilia, as measured over a period of 4 weeks on an annual basis, using the visual analog scale (VAS) | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The VAS assesses the pain using a scale of 0 (no pain) to 10 (unbearable pain).
  During screening visit and on an annual basis, the investigators shall ask participants to rate the average level of chronic pain associated with hemophilia over the period of 4 weeks prior to visit date using the VAS.
Acute pain associated with hemophilia, as measured with individual bleeding episodes, using the visual analog scale (VAS) | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  The VAS assesses the pain using a scale of 0 (no pain) to 10 (unbearable pain).
  Participants will be asked to provide ratings on level of acute pain associated with each bleeding episode using the VAS. The VAS scores will be recorded in the participant diary.
Number of days lost from school or work due to bleeding episodes | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
Modalities of switching from a standard FVIII product to rAHF-PEG - 1 | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  Difference in number of weekly prophylactic infusions between previous regimen and rAHF-PEG
Modalities of switching from a standard FVIII product to rAHF-PEG - 2 | Enrollment visit; Screening visit; Annual/Interval visits: - Up to 8 years if rAHF-PFM alone - Up to 8 years if rAHF-PEG alone with minimum follow up of 4 years - Up to approx. 12 years rAHF-PFM and switched to rAHF-PEG; Termination visit
  Difference in number of weekly doses between previous regimen and rAHFPEG
Incidence of Inhibitors in Previously Treated Patients (PTPs) with Factor VIII (FVIII) Levels Lesser than (<)1%, Lesser Than or Equal to (<=) 2%, and <= 5% without history of inhibitor | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
Incidence of Inhibitors in Previously Treated Patients (PTPs) with Factor VIII (FVIII) Levels <1%, <=2%, and <= 5% with history of inhibitor | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
Incidence of Inhibitors in Previously Untreated Patient (PUPs) and Minimally Treated Patients (MTPs) with Factor VIII (FVIII) Levels <1%, <=2%, and <= 5% | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
Incidence of therapy-related serious adverse events | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
Incidence of therapy-related non-serious adverse events | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
Incidence of inhibitors after switching to rAHF-PEG | Throughout the study period of up to approximately: 8 years (rAHF-PFM alone), or 12 years (rAHF-PEG alone or after receiving rAHF-PFM)
  Incidence of inhibitors after switching to rAHF-PEG in the same subgroups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (110):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - South Metropolitan Health Service trading as Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Landes Frauen und Kinderklinik Linz (LFKK Linz), Linz
  - Kepler Universitätsklinikum Klinik für Kinder-und Jugendheilkunde, Linz
  - Medizinische Universitaet Wien, Vienna
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Brazil (9):
  - Hemoce - Ce, Fortaleza, Ceará
  - Hemocentro do Espírito Santo, Vitória, Espírito Santo
  - Hemepar - Pr, Curitiba, Paraná
  - Hemorgs - Rs, Porto Alegre, Parthenon
  - Fundação HEMOPA, Belém, Pará
  - Hemocentro da UNICAMP, Campinas, São Paulo
  - Hemocentro Ribeirão Preto - SP, Ribeirão Preto, São Paulo
  - Hemorio - Rj, Rio de Janeiro
  - Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Canada (6):
  - Stollery Children's Hospital, University of Alberta, Edmonton, Alberta
  - The Moncton City Hospital, Moncton, New Brunswick
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - St-Michael's Hospital, Toronto, Ontario
  - Sick Kids Hospital, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (9):
  - Shenzhen Children's Hospital, Shenzhen, Futian
  - Nanfang Hospital Affiliated to Nanfang Medical University, Guangzhou, Guangdong
  - Institute of Hematology, Blood Disease Hospital, PUMC&CAMS, Tianjin, Heping
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Blood Center of Shandong Province, Jinan, Shandong
  - Beijing Children's Hospital Affiliated to Capital University of Medical Sciences, Beijing
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Shenzhen Second People's Hospital, Shenzhen
- Colombia (3):
  - IPS FUSA SAS Centro Integral de Coagulacion, Atlántico
  - Integral Solutions SD SAS, Bogotá
  - Fundación Oftalmológica de Santander FOSCAL, Floridablanca
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Ostrava, Oddělení dětské hematologie a hematoonkologie, Ostrava
  - Fakultní nemocnice Ostrava, Ostrava
  - Fakultní nemocnice v Motole, Prague
- Rigshospitalet, Copenhagen, Denmark
- France (13):
  - "Hôpital Morvan CHRU de Brest", Brest
  - CHU Côte de Nacre - CRTH, Caen
  - Centre Hospitalier Générale - CTH, Chambéry
  - CTRH - CHU Bocage, Dijon
  - Hôpital André Mignot, Le Chesnay
  - Hôpital de la Mère et de l'Enfant - CHU de LIMOGES, Limoges
  - CHRU Hôtel Dieu - CRTH, Nantes
  - Hôpital Cochin, Paris
  - CHU de Reims Hôpital Maison Blanche - CRTH, Reims
  - Centre Régional de Traitement de l'Hémophilie et des Maladies hémorragiques. CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHRU Charles Nicolle, Rouen
  - CIC, Saint-Priest-en-Jarez
  - CHRU Purpan CRTH - Pavillon Sénac, Toulouse
- Greece (3):
  - Aghia Sofia Children's Hospital, Goudi, Athens
  - Laikon General Hospital, Goudi, Athens
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Hungary (5):
  - Heim Pál Gyermekkórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Mohács City Hospital, Mohács
  - Jósa András County Hospital, Nyíregyháza
  - Markusovszky Hospital, Szombathely
- Italy (16):
  - Azienda Ospedaliera Policlinico Consorziale Di Bari, Bari
  - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Vittorio Emanuele, Ferrarotto, S. Bambino, Catania
  - Ospedale Pugliese -Ciaccio, Catanzaro
  - Az. Osp. Univ. Careggi, Florence
  - Ospedale di Macerata, Macerata
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera di Padova Clinica Medica II, Padua
  - AOUP P. Giaccone, Palermo
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Università degli studi di Roma "La Sapienza", Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Policlinico Universitario Gemelli, Roma
  - Centro Emofilia e Coagulopatie Rare, Scorrano
  - Ospedale Molinette, Torino
- Norway (2):
  - Rikshospitalet, Oslo
  - Rikshospitalet, Oslo University Hospital, Oslo
- Poland (4):
  - Szpital Uniwersytecki nr 1 im. dr Andrzeja Jurasza, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Gdansk
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wrocławiu, Wroclaw
- Portugal (4):
  - Hospital do Divino Espírito Santo, Ponta Delgada, Azores
  - Centro Hospitalar e Universitade de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte Hospital de Sta. Maria, Lisbon
  - Centro Hospitalar de São João, E.P.E., Porto
- Russia (5):
  - SBHI Chelyabinsk Regional Children's Clinical Hospital, Chelyabinsk
  - Federal State Budget Institution "Hematology Research Center" of Ministry of Healthcare of Russian Federation, Moscow
  - SBHI of the Republic of Kareliya Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - State Budget Healthcare Institution of Saint-Petersburg "City polyclinic #37", Saint Petersburg
  - Clinics of FSBEI High Education Samara SMU of MoH of Russia, Samara
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (4):
  - Hospital Teresa Herrera-Materno Infantil, A Coruña
  - Hospital Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitari Vall d'Hebron (HUVH), Barcelona
  - Hospital Universitario Son Espases, Palma de Mallorca
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Kliniska studier i Sverige - Forum Söder, Malmo
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (8):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - FMH Kinder und Jugendmedizin, im Wabern-Zentrum, Wabern
  - Kinderspital Zürich, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Cambridge University Hospital NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - East Kent Hospitals University Foundation Trust, Kent & Canterbury Hospital, Canterbury
  - Great Ormond Street Hospital for Children NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ozelo MC, Hermans C, Carcao M, Guillet B, Gu J, Guerra R, Tang L, Khair K. The effectiveness and safety of octocog alfa in patients with hemophilia A: up to 7-year follow-up of the real-world AHEAD international study. Ther Adv Hematol. 2024 Feb 15;15:20406207231218624. doi: 10.1177/20406207231218624. eCollection 2024. PMID 38371314
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc24db2bf003ab45765